CLINICAL TRIAL: NCT04943731
Title: Changes in Pulmonary Outcomes as a Result of Implementing a Day and Night Regimen With Heat and Moisture Exchangers (HMEs) and Their Attachments
Brief Title: Day/Night Regimen With Provox Life Heat and Moisture Exchangers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: Princess Alexandra Hospital, Brisbane, Australia (Other); Royal Brisbane and Women's Hospital (Other Government); Prince of Wales Hospital, Sydney (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HREC/2021/QMS/74792
Record Dates: First submitted 2021-06-07; First posted 2021-06-29 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Laryngectomy
Keywords: Pulmonary rehabilitation; Heat and Moisture Exchangers

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, two-phase clinical study. The end of Phase 1 serves as the baseline for Phase 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Provox Life™ (Other): Phase 1: Provox Life™. Like-for-like transition from Provox (or other brand) to Provox Life™ under guidance from Speech Pathologist who will assess when the participant is ready to commence the 6 week study observation period.
  Phase 2: Provox Life™ with Day/Night regimen. Establishment of optimal day/night routine under guidance of Speech Pathologist who will assess when the participant is ready to commence the 6 week observation period.
  Interventions: Device: Provox Life

INTERVENTIONS:
Device: Provox Life — Phase 1: Like for like transition, Phase 2: Provox Life day/night regimen

SUMMARY:
Purpose and Aim: This research is about patients who have had a total laryngectomy, trialing a new range of Heat and Moisture Exchangers (HMEs) - referred to as the "Provox Life™ range of HMEs". The main purpose of this study is to find out if participants experience any differences in the amount of coughing and mucus problems when using the new range of Provox Life™ HMEs (and attachment devices) following an optimal Day/Night regimen. The study is sponsored by Atos Medical.

Study Design: Participants will use the new Provox Life™ HME range and their attachments during two (2) observation phases (Phase 1, Phase 2). In Phase 1 (6 week study phase), participants will use the new Provox Life™ HMEs in a similar way as they currently use their existing HME devices. In the Phase 2 (6 week study phase), they will use the Provox Life™ HME devices following an optimal Day/Night regimen - with the aim to achieve the best possible humidification at all times. Prior to each study phase, participants will meet with their speech pathologist to learn about the new devices and how to use them. Once comfortable using them they will commence each observation phase.

Data Collection: Experiences using their existing HMEs (prior to study) and then using the new HMEs in Phase 1 and Phase 2 will be collected via a series of questionnaires. These will be completed 5 times in total - at baseline before Phase 1 starts, and then at both week 2 and week 6 of Phase 1 and 2. Questionnaires relate to their use of the HMEs, coughing and mucus problems, skin integrity, overall experiences of using the new devices and any impacts on sleep and quality of life. Participants will complete some of the questionnaires at home (approx. 30mins) and the others during an interview session with one of the study team (approx. 30mins). The interview session can be conducted via telephone, videoconferencing or in person - depending on the patients preferences and any COVID restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Total laryngectomy, irrespective of pharynx reconstruction method
* 18 years or older
* HME user
* Longer than 3 months after total laryngectomy
* Longer than 6 weeks after postoperative radiotherapy

Exclusion Criteria:

* Current day/night routine with Provox Luna
* Daily use of Provox Micron HMEF
* Medical problems prohibiting the use of HME
* Active recurrent or metastatic disease (medical deterioration)
* Recent pulmonary infections/unstable pulmonary condition
* Reduced mobility of arms and/or hands, unable to insert or remove an HME
* Unable to understand the Participant Information and/or unable to give Informed Consent
* Insufficient cognitive ability to manage HME or adhesive use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in COUS score of CASA-Q | Change from End of Phase 1 (week 6) to End of Phase 2 (week 12)
  Cough Symptoms (COUS) assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q). Score between 0 and 100, with higher scores meaning less symptoms and less impact.
Change COUI scores of CASA-Q | Change from End of Phase 1 (week 6) to End of Phase 2 (week 12)
  Cough Impact (COUI) assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q). Score between 0 and 100, with higher scores meaning less symptoms and less impact.

SECONDARY OUTCOMES:
Change in SPUS score of CASA-Q | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Sputum Symptoms (SPUS) domains of the CASA-Q. Score between 0 and 100, with higher scores meaning less symptoms and less impact.
Change in SPUI score of CASA-Q | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Sputum Impact (SPUI) domains of the CASA-Q. Score between 0 and 100, with higher scores meaning less symptoms and less impact.
Change in COUS scores of CASA-Q | Baseline, Phase 1 (2 weeks), and Phase 2 (2 weeks)
  Cough Symptoms (COUS) assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q). Score between 0 and 100, with higher scores meaning less symptoms and less impact.
Change in COUI scores of CASA-Q | Baseline, Phase 1 (2 weeks), and Phase 2 (2 weeks)
  CCough Impact (COUI) assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q). Score between 0 and 100, with higher scores meaning less symptoms and less impact.
Number of forced mucus expectorations per 24 hours | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Patient reported, recorded by tally sheeting
Number of involuntary coughs per 24 hours | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Patient reported, recorded by tally sheeting
Quality of Life by EQ-5D-5L | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  patient reported, the descriptive system assesses health in five dimensions, from which a health state index score is calculated, range from 0 to 1, with higher scores indicatinghigher health utility
Questionnaire for Skin Integrity | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Patient reported
Jenkins sleep evaluation questionnaire | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Patient reported to assess sleep quality. Score between 0 and 20, with higher score the more sleep disturbances
Questionnaire to assess Shortness of Breath | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  from Ackerstaff et al., 1993
Questionnaire to adjustment to Day/Night regimen | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Study specific questionnaire to describe patients adjustment to Day/Night regimen
Consumption of medical devices (Number of devices used) | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Number of devices used, by use of patient diary recoding number of devices used
Study-specific questionnaire to assess number of complications and medical treatments | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  Study specific questionnaire to record complications and consumption of medications, diagnostics, treatment, medical care, medical transportation, sick leave
Study-specific questionnaire to assess patients satisfaction | Baseline, Phase 1 (2 weeks, 6 weeks), Phase 2 (2 weeks, 6 weeks)
  patient satisfaction with devices and regimen

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Ward, PhD, Principal Investigator — Centre for functioning and Health Research, Metro South Hospital and Health Service
Locations (3):
- Australia (3):
  - Prince of Wales Hospital, NSW, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ward EC, Hancock K, Boxall J, Burns CL, Spurgin AL, Lehn B, Hoey J, Robinson R, Coleman A. Post-laryngectomy pulmonary and related symptom changes following adoption of an optimal day-and-night heat and moisture exchanger (HME) regimen. Head Neck. 2023 Apr;45(4):939-951. doi: 10.1002/hed.27323. Epub 2023 Feb 20. PMID 36808179